CLINICAL TRIAL: NCT06499298
Title: Retrospective Evaluation of Nivolumab in Adjuvant Esophageal Cancer/Gastroesophageal Junction Cancer: A Non-interventional Study in China
Brief Title: Retrospective Evaluation of Nivolumab in Adjuvant Esophageal Cancer/Gastroesophageal Junction Cancer
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1428
Record Dates: First submitted 2024-06-21; First posted 2024-07-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer; Gastroesophageal Junction Cancer
Keywords: Esophageal Cancer (EC); Gastroesophageal Junction Cancer (GEJC)
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants receiving adjuvant nivolumab
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — As per product label, as prescribed by treating physician

SUMMARY:
The purpose of this study is to describe the real-world effectiveness and patterns of use of adjuvant nivolumab in adult participants with Stage II/III Esophageal Cancer/Gastroesophageal Junction Cancer (EC/GEJC) in China.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older at the index date
* All patients must have Stage II or Stage III carcinoma of the esophagus or gastroesophageal junction and have histologically or cytologically confirmed predominant adenocarcinoma or squamous cell carcinoma esophageal or gastroesophageal junction cancer at the time of initial diagnosis.
* Participants initiated nivolumab in adjuvant Esophageal Cancer (EC) or gastroesophageal junction cancer (GEJC) treatment within the index window.

Exclusion Criteria:

* Participation in a clinical trial of an investigational drug concurrently during the adjuvant nivolumab treatment.
* From the date of diagnosis of EC or GJEC to data end period, patients were diagnosed with a primary diagnosis of a cancer other than EC or GJEC that requires systemic or other treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult participants from China with Stage II/III Esophageal Cancer/Gastroesophageal Junction Cancer (EC/GEJC) who initiated nivolumab treatment in routine clinical practice between June 27, 2022 and October 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Participant disease-free survival (DFS) | Up to 1 year

SECONDARY OUTCOMES:
Participant socio-demographics | Baseline and up to 1 year
Date of tumor initial diagnosis | Baseline
Tumor location at initial diagnosis | Baseline
Tumor histology at initial diagnosis | Baseline
Resected tumor margins status | Baseline
  Negative (clear), positive (involved), close margins
Eastern Cooperative Oncology Group (ECOG) performance status | Baseline and up to 1 year
Pathological lymph-node status | Baseline and up to 1 year
Pathological tumor status | Baseline and up to 1 year
Participant biomarkers (if available) | Baseline and up to 1 year
  Including PD-L1 expression, HER2 status, Epstein-Barr virus positivity, tumor metastasis
Participant outcomes after nivolumab treatment | Baseline and up to 1 year
  Including disease stage, recurrence, disease progression, medical imaging test result, and death information
Participant medical history | Baseline and up to 1 year
Participant cancer treatment history | Baseline
Esophageal Cancer (EC) or gastroesophageal junction cancer (GEJC) stage at nivolumab treatment initiation | Day 1
Indication for nivolumab treatment | Day 1
Nivolumab treatment duration | Up to 1 year
Time from surgery to nivolumab initiation | Day 1
Nivolumab treatment regimen | Up to 1 year
Participant concomitant treatment(s) | Baseline and up to 1 year
Participant systemic treatment(s) | Up to 1 year
Date of nivolumab treatment completion/discontinuation | Up to 1 year
Reasons for treatment discontinuation/cessation | Up to 1 year
Subsequent treatment after nivolumab discontinuation | Up to 1 year
Time to next treatment (TTNT) | Up to 1 year
Nivolumab treatment modifications in relation to the management of adverse events (AE) | Up to 1 year
Participant distant metastasis-free survival (DMFS) | Up to 1 year
Participant distant metastasis-free survival (DMFS) rates | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts